CLINICAL TRIAL: NCT06901167
Title: Evaluation of a Region-wide Residential In-Reach (RIR) Program in Regional and Rural Health Services: A Stepped-wedge Trial
Brief Title: Evaluation of a Residential In-Reach Program in Regional and Rural Australia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Monash University (Other)
Collaborators: Deakin University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HREC/112397/GHSJOG-2025-462490
Record Dates: First submitted 2025-03-04; First posted 2025-03-28 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-03

CONDITIONS: Aged; Acute Disease
Keywords: stepped-wedge trial; residential aged care home; residential in reach; hospital avoidance
MeSH Terms: conditions — Acute Disease

STUDY DESIGN:
Intervention Model Description: This will be a stepped-wedge trial, in which all enrolled facilities and participants will receive the same intervention, but the intervention roll-out will be conducted in a sequential manner based on a randomised order. During the 14 months of the trial, all facilities and participants will receive the same intervention, but for different lengths of time depending on the randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Residential-in-reach (Experimental): All enrolled residential aged care homes will be able to access the residential-in-reach (RIR) program intervention. The RIR program provides a consultation service from a central hospital to an aged care facility in the Grampians region in the state of Victoria, Australia. Aged care staff will make a telehealth referral to central hub, where a nurse practitioner will triage the patient and make recommendations (for example, monitor resident condition, more examples: comprehensive assessment for unwell residents, liaison with the General Practitioners for diagnosis and treatment plan, provide education and support to staff) or further referrals (for example, refer to geriatrician or call an ambulance).
  Interventions: Other: Residential In-Reach Program

INTERVENTIONS:
Other: Residential In-Reach Program — All enrolled residential aged care homes will be able to access the residential-in-reach (RIR) program intervention. The RIR program provides a consultation service from a central hospital to an aged care facility in the Grampians region in the state of Victoria, Australia. Aged care staff will make a telehealth referral to central hub, where a nurse practitioner will triage the patient and make recommendations (for example, monitor resident condition, more examples: comprehensive assessment for unwell residents, liaison with the General Practitioners for diagnosis and treatment plan, provide education and support to staff) or further referrals (for example, refer to geriatrician or call an ambulance).

SUMMARY:
Residential In-Reach (RIR) programs are designed to provide responsive care for residents in residential aged care homes (RACH) with the aim of avoiding unnecessary hospital transfers. The evidence for their clinical and cost-effectiveness and implementation has been established in urban settings, but there is a small amount of low-quality evidence for rural and regional settings. The Grampians Region Health Service Partnership Resi-In-Reach Redesign Committee will be implementing a new RIR program to be offered to all RACHs in the Grampians region, this project aims to evaluate the clinical and cost-effectiveness of this program, and its implementation in the rural and regional setting. A stepped-wedge trial will be conducted so that as the RIR program is gradually rolled-out across the region, outcomes can be compared in the same facilities across time and between different facilities. The primary outcome measure will be presentation to emergency departments and urgent care centres, and data will also be collected on other clinical outcomes and barriers and enablers of implementing the program. It is anticipated that there will be a reduction in hospital presentations, and a range of barriers and enablers unique to the rural and regional setting will emerge.

ELIGIBILITY:
Inclusion Criteria:

* Health services that have emergency departments and/or emergency care centres that admit residents from residential aged care homes (RACH)
* RACHs that do not currently have access to RIR programs
* health service staff who have been involved with the set-up and delivery of the RIR program,
* RACH staff who have experience of or accessing the RIR service for residents at least once,
* residents living at a RACH who has experienced receiving medical care from the RIR program and can provide informed consent, or a family member of the resident,
* general practitioners whose case load includes residents from RACHs.

Exclusion Criteria:

• RACHs that already have access to a RIR program will be excluded

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of presentations from residential aged care homes to emergency departments and emergency care centres | From enrolment to the end of the trial for 14 months
  Primary clinical effectiveness outcome
  Collection schedule:
  * Once at the end of the evaluation
  * At the level of each residential aged care home presentation to hospital each month Collection approach: Extraction from hospital records and extraction from residential aged care home systems

SECONDARY OUTCOMES:
Days spent in hospital by aged care home resident | From enrolment to the end of the trial for 14 months
  Secondary clinical effectiveness outcome
  Collection schedule:
  * Once at the end of the evaluation
  * At the level of each residential aged care home presentation to hospital each month Collection approach: Extraction from hospital records and extraction from residential aged care home systems
Location of mortality in hospital | From enrolment to the end of the trial for 14 months
  Secondary clinical effectiveness outcome
  Collection schedule:
  * Once at the end of the evaluation
  * At the level of each residential aged care home presentation to hospital each month Collection approach: Extraction from hospital records and extraction from residential aged care home systems
Number of barriers to residential-in-reach program implementation | From enrolment to 1 month after the end of the trial, for 15 months
  Secondary implementation outcome - collected once via semi-structured interviews with key stakeholders (health service staff, residential aged care home staff).
Number of enablers to residential-in-reach program implementation | From enrolment to 1 month after the end of the trial, for 15 months
  Secondary implementation outcome - collected once via semi-structured interviews with key stakeholders (health service staff, residential aged care home staff).
Stakeholder reported feasibility of the residential-in-reach program implementation | From enrolment to 1 month after the end of the trial, for 15 months
  Secondary implementation outcome - collected once via semi-structured interviews with key stakeholders (health service staff, residential aged care home staff).
Stakeholder reported acceptability of the residential in-reach program | From enrolment to the end of the trial for 14 months
  Secondary implementation outcome - collected via semi-structured interviews with key stakeholders (health service staff, residential aged care home staff, general practitioners, aged care home residents) after occasions of service on a monthly basis.
Stakeholder reported appropriateness of the residential in-reach program | From enrolment to the end of the trial for 14 months
  Secondary implementation outcome - collected via semi-structured interviews with key stakeholders (health service staff, residential aged care home staff, general practitioners, aged care home residents) after occasions of service on a monthly basis.
Number of aged care staff who attend education sessions for the use of the residential in-reach program | From enrolment to the end of the trial for 14 months
  Secondary implementation outcome - recorded attendance of education sessions for residential aged care home staff for the use of the residential in-reach program.
Number of adaptations made to the residential in-reach program | From enrolment to the end of the trial fo
  Secondary implementation outcome - documented adaptations made to the program during the trial period.

OTHER OUTCOMES:
Number of times the residential in-reach program is utilised | From enrolment to the end of the trial for 14 months
  Cost-effectiveness outcome: number of times the RACHs enrolled in this trial utilises the residential in-reach program, both in-person and via telehealth.
  Collection schedule:
  * Once at the end of the evaluation
  * At the level of each residential aged care home each month Collection approach: Extraction from hospital records
Number of times the Victorian Virtual Emergency Department is utilised | From enrolment to the end of the trial for 14 months
  Cost-effectiveness outcome: number of times the RACHs enrolled in this trial uses the Victorian Virtual Emergency Department.
  Collection schedule:
  * Once at the end of the evaluation
  * At the level of each residential aged care home each month Collection approach: Extraction from residential aged care home records
Number of times that the general practitioner is utilised | From enrolment to the end of the trial for 14 months
  Cost-effectiveness outcome: number of times that the RACHs enrolled in this trial consults the general practitioner, both in-person and via telehealth, including in and out of hours consultations.
  Collection schedule:
  * Once at the end of the evaluation
  * At the level of each residential aged care home each month Collection approach: Extraction from residential aged care home records
Number of calls to Ambulance Victoria | From enrolment to the end of the trial for 14 months
  Cost-effectiveness outcome: number of times the RACHs enrolled in this trial calls an ambulance for their residents.
  Collection schedule:
  * Once at the end of the evaluation
  * At the level of each residential aged care home each month Collection approach: Extraction from residential aged care home records and Ambulance Victoria records
Number of transfers to hospital via Ambulance Victoria | From enrolment to the end of the trial for 14 months
  Cost-effectiveness outcome: number of times that Ambulance Victoria transfers a resident from one of the RACHs enrolled in this trial to hospital.
  Collection schedule:
  * Once at the end of the evaluation
  * At the level of each residential aged care home each month Collection approach: Extraction from residential aged care home records and Ambulance Victoria records

CONTACTS AND LOCATIONS:
Overall Officials: Terry Haines, Principal Investigator — Monash University
Locations (8):
- Australia (8):
  - East Grampians Health Service, Ararat, Victoria
  - Grampians Health, Ballarat, Victoria
  - Beaufort and Skipton Health Service, Beaufort, Victoria
  - Central Highlands Rural Health, Daylesford, Victoria
  - Maryborough District Health Service, Maryborough, Victoria
  - West Wimmera Health Service, Nhill, Victoria
  - East Wimmera Health Service, Saint Arnaud, Victoria
  - Rural Northwest Health, Warracknabeal, Victoria

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be analysed and reported on. Planned data management involves analysis and reporting of aggregated data from all participants from all sites.

REFERENCES:
- [Background] Sunner C, Giles MT, Parker V, Dilworth S, Bantawa K, Kable A, Oldmeadow C, Foureur M. PACE-IT study protocol: a stepped wedge cluster randomised controlled trial evaluating the implementation of telehealth visual assessment in emergency care for people living in residential aged-care facilities. BMC Health Serv Res. 2020 Jul 20;20(1):672. doi: 10.1186/s12913-020-05539-1. PMID 32690008
- [Background] Sunner C, Giles MT, Kable A, Foureur M. Experiences of nurses working in RACFs and EDs utilising visual telehealth consultation to assess the need for RACF resident transfer to ED: A qualitative descriptive study. J Clin Nurs. 2023 Aug;32(15-16):4694-4709. doi: 10.1111/jocn.16529. Epub 2022 Sep 8. PMID 36081333
- [Background] Lukin B, Fan LJ, Zhao JZ, Sun JD, Dingle K, Purtill R, Tapp S, Hou XY. Emergency department use among patients from residential aged care facilities under a Hospital in the Nursing Home scheme in public hospitals in Queensland Australia. World J Emerg Med. 2016;7(3):183-90. doi: 10.5847/wjem.j.1920-8642.2016.03.004. PMID 27547277
- [Background] Hullick C, Conway J, Hall A, Murdoch W, Cole J, Hewitt J, Oldmeadow C, Attia J. Video-telehealth to support clinical assessment and management of acutely unwell older people in Residential Aged Care: a pre-post intervention study. BMC Geriatr. 2022 Jan 10;22(1):40. doi: 10.1186/s12877-021-02703-y. PMID 35012480
- [Background] Haines TP, Palmer AJ, Tierney P, Si L, Robinson AL. A new model of care and in-house general practitioners for residential aged care facilities: a stepped wedge, cluster randomised trial. Med J Aust. 2020 May;212(9):409-415. doi: 10.5694/mja2.50565. Epub 2020 Apr 1. PMID 32237279
- [Background] Chambers D, Cantrell A, Preston L, Marincowitz C, Wright L, Conroy S, Lee Gordon A. Reducing unplanned hospital admissions from care homes: a systematic review. Health Soc Care Deliv Res. 2023 Oct;11(18):1-130. doi: 10.3310/KLPW6338. PMID 37916580